CLINICAL TRIAL: NCT06321731
Title: Observational Retrospective Study To Describe Characteristics And Evaluate Real-World Outcomes in COPD Patients Initiating Trixeo Aerosphere (Budesonide/Glycopyrronium Bromide/Formoterol Fumarate) in Spain
Brief Title: Real-World Outcomes in COPD Patients Starting Trixeo (Budesonide/Glycopyrronium/Formoterol) in Spain.
Acronym: ORESTES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00096
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients initiating BGF: COPD patients ≥40 years old initiating BGF (budesonide/glycopyrronium bromide/formoterol fumarate) at least 12 months before start of data collection.

SUMMARY:
The aim of the ORESTES study is to describe the characteristics of the COPD patients initiating Trixeo (BGF -budesonide/glycopyrronium/formoterol) in Spain and to assess their real-world outcomes up to 12 months afterwards.

For that purpose,a descriptive, observational, multi-centre, longitudinal, retrospective cohort study involving ~20 Spanish centres and aiming to include between 500 and 700 patients, has been designed.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by irreversible airflow obstruction, and it is a significant global health concern. According to the World Health Organization (WHO) COPD is the third leading cause of death worldwide, causing 3.23 million deaths in 2019. In Spain, around 12% of the population over 40 (approximately 2.2 million people) suffer from COPD, with an 11% mortality rate following hospitalization for a COPD exacerbation.

COPD exacerbations, associated with reduced quality of life, increased healthcare utilization, and substantial mortality, are more likely to recur in patients who have experienced one moderate or severe exacerbation. Traditionally, long-term bronchodilator therapy has been the primary pharmaceutical approach, including β2 agonists, anticholinergics, and inhaled corticosteroids (ICS). Triple therapy (TT), combining a long-acting β2 agonist (LABA), long-acting anticholinergic (LAMA), and ICS, is recommended for patients with persistent exacerbations.

Trixeo Aerosphere®, a fixed-dose combination of ICS/LABA/LAMA (budesonide/glycopyrronium bromide/formoterol fumarate, hereafter BGF) in a single inhaler, was approved in the European Union in December 2020 and marketed in Spain from February 2022. The Phase III ETHOS trial demonstrated significant reductions in moderate to severe exacerbations, improved quality of life, and lung function compared to dual therapies.

To assess real-world outcomes of patients initiating BGF in Spain, the ORESTES study has been designed.

The study primary objective is to describe the occurrence and severity of exacerbations of COPD-diagnosed patients receiving BGF from treatment initiation to end of treatment, loss to follow-up, death or up to 12 months of treatment.

The study secondary objectives are:

1. To describe the demographic and clinical profile of patients at the moment of BGF initiation.
2. To describe other patients' clinical outcomes (apart from exacerbations), treatment outcomes and healthcare resource utilisation (HCRU) after initiation of BGF.

The study exploratory objectives are:

1. To describe severe cardiovascular (CV)-related outcomes after initiation of BGF.
2. To describe the mortality after initiation of BGF.

Descriptive, observational multi-centre, longitudinal, retrospective cohort study aiming to include adult patients aged 40 years or older diagnosed with COPD and who initiated BGF at least 12 months before inclusion.

The study observation period runs from 12 months prior to the start of BGF, defined as the index date, until the censoring date, i.e., the earliest of BGF treatment discontinuation, loss to follow-up, death or maximum of 12 months after index date.

This study is based exclusively on secondary data collection from outpatient electronic medical records (EMRs). Therefore, it will rely on already existing data from patients by the time of data collection.

The study will include 500-700 patients from approximately 20 hospitals in Spain.

ELIGIBILITY:
Inclusion Criteria:

1 .Patient diagnosed with COPD confirmed by spirometry (postbronchodilator FEV1/FVC<0.7).

2. Patients treated with BGF initiated at least 12 months before start of data collection.

3. Patients with information available at least 12 months before BGF initiation.

4. Adult patients aged ≥40 years old at index date.

Exclusion Criteria:

1. Subjects with BGF treatment not intended for COPD (e.g., intended for asthma).
2. Subject participated in a clinical trial during the study data observation period.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 500-700 COPD patients who started BGF treatment at least 12 months before start of data collection, and from approximately 20 hospitals in Spain.
Sampling Method: Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Annualized rate of exacerbations after BGF initiation | Up to 12 months
  Annualized rate (total number of exacerbations divided by the total number of person years) of exacerbations occurred during the study data observation period after BGF initiation, overall and classified by severity (severe and moderate).

SECONDARY OUTCOMES:
Demographic and clinical profile of patients initiating BGF. | Index date (BGF initiation) and baseline (previous 12 months)
  Patient demographics, comorbidities, clinical characteristics related to COPD and other respiratory-related variables such as lung function and dyspnoea, the presence of eosinophils, exacerbations, medication used for COPD, including OCS and rescue medication, and the healthcare resource use (HCRU).
Lung Function after BGF initiation | Up to 12 months
  Measured by forced expiratory volume at first second (FEV1), FEV1 of the predicted %, forced vital capacity (FVC) volume and % FEV1/FVC
Eosinophils count after BGF initiation | Up to 12 months
  Counts in cells/µL
Persistence to treatment (BGF) | Up to 12 months
  Duration time from initiation to discontinuation of treatment
Need for rescue medication after BGF initiation | Up to 12 months
  Number of uses per year and time to first use
Use of oral corticosteroids (OCS) after BGF initiation | Up to 12 months
  Frequency and cumulative dosage (mg)
HCRUs related to COPD after BGF initiation | Up to 12 months
  Annualized rate of specialist visits, general practitioner (GP) visits, ER admissions and hospitalizations (along with duration)

OTHER OUTCOMES:
Annualized rate of severe cardiovascular (CV)-related outcomes after initiation of BGF. | Up to 12 months
  CV-related outcomes occurred after treatment initiation: tachyarrhythmias, heart failure (HF), and myocardial infarction (MI) and stroke, measured by the number of events per year and severity, and as a time to event variable, from treatment initiation.
Mortality (% and time to event) after BGF initiation | Up to 12 months
  2. Patient's mortality will be measured by percentage of deaths and reason of deaths (CV-related, respiratory-related, other) and as a time to event variable, from treatment onset to occurrence of death.

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Lleida
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza

REFERENCES:
- [Derived] Figueira-Goncalves JM, Alcazar-Navarrete B, Casitas-Mateo R, Gonzalez J, Gotera-Rivera CM, Herrejon-Silvestre A, Margallo-Iribarnegaray J, Martin-Lana M, Pallares-Sanmartin A, Pascual-Guardia S, Saura-Vinuesa A, Corregidor-Garcia C, Fitas E, Sanchez-Covisa J. Real-World Outcomes in Patients with COPD Initiating Budesonide/Glycopyrronium/Formoterol Fumarate Dihydrate After Dual and Triple Therapy in Spain: A Sub-Study of the ORESTES Study. Pulm Ther. 2026 Jan 19. doi: 10.1007/s41030-026-00341-6. Online ahead of print. PMID 41553424
- [Derived] Alcazar-Navarrete B, Figueira-Goncalves JM, Corregidor-Garcia C, Fitas E, Sanchez-Covisa J; ORESTES group. Real-World Outcomes in Patients with COPD Initiating Budesonide/Glycopyrronium/Formoterol Fumarate Dehydrate in Spain: ORESTES Study. Adv Ther. 2025 Nov;42(11):5708-5726. doi: 10.1007/s12325-025-03361-x. Epub 2025 Sep 22. PMID 40982160
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00096&attachmentIdentifier=4cb3deaa-8cd0-4117-aa74-24fa21805fac&fileName=Redacted_CSR_Synopsis_D5980R00096.pdf&versionIdentifier=